CLINICAL TRIAL: NCT02049164
Title: A Randomized, Double-blind, Placebo-controlled, Forced Titration, Dose-ranging Study of AR08 in the Treatment of Vasomotor Symptoms (VMS) in Menopausal Females: A Proof-of-Concept Study
Brief Title: Safety and Efficacy Study of AR08 for the Treatment of Vasomotor Symptoms (VMS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopping criteria met with regards to vital sign measurements post dose.
Sponsor: Arbor Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR08.100
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-11

CONDITIONS: Vasomotor Symptoms (VMS)
Keywords: AR08, Vasomotor Symptoms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AR08 0.5 mg/day (Experimental): AR08 QD oral dosing for 14 weeks
  Interventions: Drug: AR08
- AR08 1.0 mg/day (Experimental): AR08 QD oral dosing for 14 weeks
  Interventions: Drug: AR08
- AR08 2.0 mg/day (Experimental): AR08 QD oral dosing for 14 weeks
  Interventions: Drug: AR08
- Placebo (Placebo Comparator): Placebo QD oral dosing for 14 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AR08
  Arms: AR08 0.5 mg/day; AR08 1.0 mg/day; AR08 2.0 mg/day
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effective dose or dose range of AR08 in the treatment of VMS in menopausal females.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy female > 40 years of age with a body mass index (BMI) ≤ 40;
2. Has undergone menopause defined as any of the following:

   At least 12 months of spontaneous amenorrhea; or At least 6 months of spontaneous amenorrhea with serum follicle-stimulating hormone (FSH) levels > 40 mIU/mL; or At least 6 weeks postsurgical bilateral oophorectomy (with or without hysterectomy);
3. Experience a minimum of 7 moderate to severe hot flushes per day or 50 moderate to severe hot flushes per week

Exclusion Criteria:

1. Resting systolic blood pressure (SBP) <110 mmHg, resting diastolic blood pressure (DBP) <50 mm Hg, or a resting heart rate (HR) <60 beats per minute while awake;
2. Subjects with pre-existing orthostatic hypotension at Screening;
3. Use of oral estrogen-, progestin-, androgen-, or selective estrogen receptor modifier (SERM) -containing drug products within 8 weeks prior to Screening; use of transdermal hormone products within 8 weeks prior to Screening; use of vaginal hormone products (rings, creams, gels) within 4 weeks prior to Screening; use of intrauterine progestins within 8 weeks prior to Screening; use of progestin implants or estrogen injectables within 3 months prior to Screening; use of estrogen pellet or progestin injectables within 6 months prior to Screening;
4. History of daily usage (at least 28 days/month) of either of the following during the month prior to initiation of Screening: Antihypertensives or Prophylactic antimigraine medications

Min Age: 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Mean change from Baseline in the frequency and severity of moderate to severe hot flashes | Weeks 4 and 12

SECONDARY OUTCOMES:
Patient Global Impression - Improvement (PGI-I) | Weeks 4, 8, and 12

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Genesis Center for Clinical Research, San Diego, California
  - Clinical Research Advantage, Inc., Colorado Springs, Colorado
  - Blue Skies Center for Women, Colorado Springs, Colorado
  - Altus Research, Lakeworth, Florida
  - OB-GYN Associates of Mid-Florida, P.A., Leesburg, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Cypress Medical Research Center, Wichita, Kansas
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Lawrence OB/Gyn Associates, Lawrenceville, New Jersey
  - Hawthorne Medical Research, Inc., Winston-Salem, North Carolina
  - Clinical Research of Philadelphia, LLC, Philadelphia, Pennsylvania
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee
  - TMC Life Research, Inc., Houston, Texas
  - Tidewater Physicians for Women, Norfolk, Virginia
  - Seattle Womens: Health, Research, Gynecology, Seattle, Washington